CLINICAL TRIAL: NCT01849055
Title: A Multiple-Dose, Dose-Escalation Study to Evaluate the Safety and Tolerability of LY3023703 in Healthy Subjects
Brief Title: A Multiple Dose Study of LY3023703 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14708; I6H-MC-MCBB (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo matching LY3023703 administered orally, once daily (QD), for 28 days
  Interventions: Drug: Placebo
- LY3023703 (Experimental): Escalating doses (2.5 milligram [mg] up to 30 mg) of LY3023703 administered orally, QD, for 28 days
  Interventions: Drug: LY3023703
- Celecoxib (Active Comparator): 400 mg celecoxib administered orally, QD, for 28 days. (Positive control.)
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: LY3023703 — Administered orally
  Arms: LY3023703
Drug: Celecoxib — Administered orally
  Arms: Celecoxib

SUMMARY:
This is a study of LY3023703 in healthy participants. The purposes of this study are to look at safety, how well the study drug is tolerated, how much of the study drug gets into the blood stream and how long it takes the body to remove the study drug. The effects of LY3023703 on blood pressure after 28 days of dosing will be studied. Information about any side effects that occur will be collected. The study is expected to last 21 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy individuals based on the history and physical examinations as determined by the investigator
* Are normotensive (defined as supine systolic blood pressure [BP] less than 140 millimeters of mercury [mm Hg] and diastolic BP less than 90 mm Hg without the use of any antihypertensives) or results that are judged to be not clinically significant by the investigator

Exclusion Criteria:

* Have presence of clinically significant active bleeding or history of bleeding diathesis at the time of screening
* Have presence of active peptic ulcer disease, gastro-intestinal (GI) bleeding, chronic gastritis, inflammatory bowel disease, or chronic diarrhea
* Have evidence of other chronic liver disease
* Have any use of nonsteroidal anti-inflammatory drugs (NSAIDs), celecoxib, aspirin, or acetaminophen (at doses greater than 1 gram per day [g/day] within 14 days of admission
* Have greater than 1 plus pretibial pitting edema or 2 plus ankle or pedal edema

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo administered by mouth (PO), once a day (QD), for 28 days
- 2.5 mg LY3023703: 2.5 milligram (mg) LY3023703 administered PO, QD, for 28 days
- 7.5 mg LY3023703: 7.5 mg LY3023703 administered PO, QD, for 28 days
- 15 mg LY3023703: 15 mg LY3023703 administered PO, QD, for 28 days
- 30 mg LY3023703: 30 mg LY3023703 administered PO, QD, for 28 days
- 400 mg Celecoxib: 400 mg celecoxib administered PO, QD, for 28 days
Period: Overall Study
Arm/Group | Placebo | 2.5 mg LY3023703 | 7.5 mg LY3023703 | 15 mg LY3023703 | 30 mg LY3023703 | 400 mg Celecoxib
Started | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 7 | 8 | 8 | 8
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo administered PO, QD, for 28 days
- 2.5 mg LY3023703: 2.5 mg LY3023703 administered PO, QD, for 28 days
- Total: Total of all reporting groups
Arm/Group | Placebo | 2.5 mg LY3023703 | 7.5 mg LY3023703 | 15 mg LY3023703 | 30 mg LY3023703 | 400 mg Celecoxib | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.8 (10.6) | 43.0 (11.7) | 37.9 (12.6) | 41.4 (10.4) | 39.0 (7.7) | 39.1 (6.8) | 39.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 0 | 1 | 1 | 7
  Male | 7 | 5 | 7 | 8 | 7 | 7 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Black/African American | 3 | 2 | 3 | 2 | 3 | 5 | 18
  Multiple | 0 | 0 | 1 | 2 | 0 | 0 | 3
  Native Hawaiian/Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 5 | 6 | 4 | 4 | 3 | 3 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 8 | 8 | 8 | 8 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of serious and all other non-serious adverse events (AE), regardless of possible study drug relatedness, is located in the Reported Adverse Events module.
Time Frame: Baseline to Study Completion (up to 74 Days)
Population: Randomized participants who reported an AE that met any of the serious criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 2.5 mg LY3023703 | 7.5 mg LY3023703 | 15 mg LY3023703 | 30 mg LY3023703 | 400 mg Celecoxib
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve [AUC(0-24)] of LY3023703
Time Frame: Post-First Dose on Days 1-28 (Time Frame: Day 1: -0.5, 1, 2, 4, 8, 12, 24 hours; Days 5, 12, 20: -0.5 hours; Day 28: -0.5, 1, 2, 4, 8, 12, 24 hours.)
Population: All randomized participants who received at least one dose of the study medication and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours•nanogram/milliliter (hr•ng/mL)
Arm/Group | 2.5 mg LY3023703 | 7.5 mg LY3023703 | 15 mg LY3023703 | 30 mg LY3023703
Number analyzed (Participants) | 8 | 8 | 8 | 8
hours•nanogram/milliliter (hr•ng/mL)
  Single Oral Dose (Day 1) | 332 (41.4) | 1140 (31.7) | 2300 (12.4) | 5290 (24.0)
  Multiple Oral Doses (Day 28): number analyzed (Participants) | 8 | 7 | 8 | 8
  Multiple Oral Doses (Day 28) | 300 (39.3) | 1340 (43.7) | 2880 (19.2) | 8520 (24.7)

3. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY3023703
Time Frame: Post first dose on Day 1 through Day 28 (Time Frame: Day 1: -0.5, 1, 2, 4, 8, 12, 24 hours; Days 5, 12, 20: -0.5 hours; Day 28: -0.5, 1, 2, 4, 8, 12, 24 hours.)
Population: All randomized participants who received at least one dose of the study medication and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 2.5 mg LY3023703 | 7.5 mg LY3023703 | 15 mg LY3023703 | 30 mg LY3023703
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL
  Single Oral Dose (Day 1) | 42.6 (25.2) | 126 (35.2) | 228 (25.6) | 556 (30.1)
  Multiple Oral Doses (Day 28): number analyzed (Participants) | 8 | 7 | 8 | 8
  Multiple Oral Doses (Day 28) | 41.9 (47.5) | 151 (47.0) | 243 (28.3) | 711 (26.2)

4. Secondary Outcome: Pharmacokinetics: Time of Maximum Concentration (Tmax) of LY3023703
Time Frame: as for outcome 3
Population: All randomly assigned participants who received at least one dose of the study medication and had evaluable PK data.
Measure: Median (Full Range); unit: Hours
Arm/Group | 2.5 mg LY3023703 | 7.5 mg LY3023703 | 15 mg LY3023703 | 30 mg LY3023703
Number analyzed (Participants) | 8 | 8 | 8 | 8
Hours
  Single Oral Dose (Day 1) | 2.01 [2.00 to 4.03] | 3.00 [2.00 to 4.00] | 4.00 [2.00 to 4.00] | 4.00 [2.00 to 4.00]
  Multiple Oral Doses (Day 28): number analyzed (Participants) | 8 | 7 | 8 | 8
  Multiple Oral Doses (Day 28) | 2.00 [1.00 to 4.00] | 2.00 [2.00 to 4.00] | 4.00 [2.00 to 4.00] | 4.00 [2.00 to 8.00]

5. Secondary Outcome: Change From Baseline to Day 27 in Blood Pressure (BP)
Description: The Day 27 change from Day -1 was analyzed by using analysis of covariance (ANCOVA) with treatment as a fixed effect and baseline Day -1 as a covariate. The treatment mean, difference to placebo, and difference to celecoxib were output with corresponding 90% confidence intervals.
Time Frame: Baseline, Day 27
Population: All randomized participants who received at least one dose of study treatment and had evaluable data.
Measure: Least Squares Mean (90% Confidence Interval); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | 2.5 mg LY3023703 | 7.5 mg LY3023703 | 15 mg LY3023703 | 30 mg LY3023703 | 400 mg Celecoxib
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
millimeters of mercury (mmHg)
  Systolic Blood Pressure (SBP) | -1.45 [-4.02 to 1.12] | -2.67 [-5.56 to 0.21] | -2.54 [-5.11 to 0.04] | -2.99 [-5.65 to -0.33] | -2.98 [-5.54 to -0.42] | -5.29 [-8.10 to -2.48]
  Diastolic Blood Pressure (DBP) | 0.28 [-1.59 to 2.14] | -0.11 [-2.03 to 1.82] | -0.83 [-2.64 to 0.98] | -0.68 [-2.62 to 1.27] | -1.22 [-3.03 to 0.59] | -2.24 [-4.10 to -0.37]
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg LY3023703; SBP; Test type: Superiority; Mean Difference (Final Values) = -1.22, 90% CI 2-sided [-4.98 to 2.54]
Statistical Analysis 2: Comparison: Placebo vs 7.5 mg LY3023703; SBP; Test type: Superiority; Mean Difference (Final Values) = -1.09, 90% CI 2-sided [-4.70 to 2.53]
Statistical Analysis 3: Comparison: Placebo vs 15 mg LY3023703; SBP; Test type: Superiority; Mean Difference (Final Values) = -1.54, 90% CI 2-sided [-5.30 to 2.22]
Statistical Analysis 4: Comparison: Placebo vs 30 mg LY3023703; SBP; Test type: Superiority; Mean Difference (Final Values) = -1.53, 90% CI 2-sided [-5.16 to 2.10]
Statistical Analysis 5: Comparison: Placebo vs 400 mg Celecoxib; SBP; Test type: Superiority; Mean Difference (Final Values) = -3.84, 90% CI 2-sided [-7.74 to 0.07]
Statistical Analysis 6: Comparison: Placebo vs 2.5 mg LY3023703; DBP; Test type: Superiority; Mean Difference (Final Values) = -0.38, 90% CI 2-sided [-2.95 to 2.18]
Statistical Analysis 7: Comparison: Placebo vs 7.5 mg LY3023703; DBP; Test type: Superiority; Mean Difference (Final Values) = -1.11, 90% CI 2-sided [-3.69 to 1.48]
Statistical Analysis 8: Comparison: Placebo vs 15 mg LY3023703; DBP; Test type: Superiority; Mean Difference (Final Values) = -0.95, 90% CI 2-sided [-3.75 to 1.85]
Statistical Analysis 9: Comparison: Placebo vs 30 mg LY3023703; DBP; Test type: Superiority; Mean Difference (Final Values) = -1.49, 90% CI 2-sided [-4.09 to 1.10]
Statistical Analysis 10: Comparison: Placebo vs 400 mg Celecoxib; DBP; Test type: Superiority; Mean Difference (Final Values) = -2.51, 90% CI 2-sided [-5.23 to 0.20]

ADVERSE EVENTS:
Arm/Group | Placebo | 2.5 mg LY3023703 | 7.5 mg LY3023703 | 15 mg LY3023703 | 30 mg LY3023703 | 400 mg Celecoxib
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 3/8 | 3/8 | 4/8 | 5/8 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=8) | 2.5 mg LY3023703 (N=8) | 7.5 mg LY3023703 (N=8) | 15 mg LY3023703 (N=8) | 30 mg LY3023703 (N=8) | 400 mg Celecoxib (N=8)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood immunoglobulin e increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 1 (2) | 1 (2) | 1 (1) | 3 (4) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0/1 (0) | 1/3 (1) | 0/1 (0) | 0/0 (0) | 0/1 (0) | 0/1 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days